CLINICAL TRIAL: NCT01805414
Title: The Effect of a Targeted Breakfast Intervention on Inpatient Glycemic Control
Brief Title: Breakfast Nutrition and Inpatient Glycemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: Pro00031605
Record Dates: First submitted 2013-02-28; First posted 2013-03-06 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2013-02

CONDITIONS: Diabetes, Type 1; Diabetes, Type 2; Cardiovascular Disease; Hyperglycemia
Keywords: inpatient diabetes; inpatient diabetes nutrition
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Cardiovascular Diseases; Hyperglycemia | interventions — Breakfast; Carbohydrates

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Breakfast (Experimental): 40-45g carbs (300-350 kcal)
  Interventions: Other: Modified Carbohydrate Breakfast
- Control Breakfast (Active Comparator): These patients received the usual hospital breakfast which contained 40-45 g carbs.
  Interventions: Other: Control Breakfast

INTERVENTIONS:
Other: Modified Carbohydrate Breakfast
  Other Names: Breakfast with 40-45g carbohydrates
  Arms: Intervention Breakfast
Other: Control Breakfast
  Other Names: 40-45g carbs
  Arms: Control Breakfast

SUMMARY:
A standard hospital meal often contains a high percentage of carbohydrates (CHO), which may not be ideal for patients with diabetes. This concern is particularly pertinent to the breakfast meal, which often contains mainly CHO. Clinical observations suggested that such diets elevate pre-lunch blood glucose (BG) values. The study team compared standard hospital "no concentrated sweets (NCS)" breakfast meals with more balanced meals. The study team hypothesized that a balanced breakfast would improve pre-lunch BG values.

This 8-week pilot study was conducted at Duke Hospital on two non-ICU cardiology wards. Ward A consisted mainly of patients with a primary diagnosis of coronary artery disease (CAD). Ward B consisted mainly of patients with a primary diagnosis of congestive heart failure (CHF). The intervention breakfast menu included 5 choices containing 40-45g of CHO. All patients on Ward A (with and without diabetes) were given the intervention breakfast for the first 4 weeks of the study, while those on Ward B received standard menus (60-75g CHO in NCS meals). After 4 weeks, the standard and intervention wards were switched. Data were collected only on patients with diabetes who were able to consume meals.

ELIGIBILITY:
Inclusion Criteria:

* Adults with cardiovascular disease who were admitted to 2 pre-specified wards at Duke Medical Center during the study period
* Diagnosis of diabetes (type 1 or 2) or newly identified hyperglycemia (blood glucose of >200 on 2 separate occasions)
* Able to consume food by mouth

Exclusion Criteria:

* Intensive care patients
* No intake by mouth (enteral, parenteral, NPO)
* Taking in nutrition supplements (Ensure, etc)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 237 (Actual)
Dates: Start 2012-09; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Relative change in Blood sugar | Pre-breakfast to pre-lunch, approximately 4 hours, daily for the study duration of 8 weeks.
  The primary outcome will be the relative change between the pre-breakfast and pre-lunch blood glucose levels after the intervention breakfast. The hypothesis is that the intervention breakfast will lead to lower pre-lunch blood sugars.
  Blood glucoses will be measured before breakfast and lunch on eligible patients. This will occur every day for the duration of the study (8 weeks).
  The relative change between the pre-breakfast and pre-lunch blood glucose will be assessed by BG2 (pre-lunch) minus BG1 (pre-breakfast).

CONTACTS AND LOCATIONS:
Overall Officials: Lillian F Lien, MD, Principal Investigator — Duke Medical Center; Kathryn J Evans, NP, Study Director — Duke Medical Center; Mark N Feinglos, MD, Study Chair — Duke Medical Center
Locations (1):
- Duke Medical Center, Durham, North Carolina, United States